CLINICAL TRIAL: NCT03078621
Title: Safety and Efficacy of Transplantation of Specific Populations of Stem Cells and Mesenchymal Stem Cells for the Treatment of Cerebral Palsy
Brief Title: Bone Marrow-Derived Stem Cell Transplantation for the Treatment of Cerebral Palsy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-CP1
Record Dates: First submitted 2017-02-25; First posted 2017-03-13 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cerebral Palsy
Keywords: stem cells
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cells (Experimental): Intravenous and Intrathecal transplantation of specific populations of purified bone marrow-derived stem cells and mesenchymal stem cells.
  Interventions: Biological: Stem Cell Therapy

INTERVENTIONS:
Biological: Stem Cell Therapy — Intravenous and Intrathecal transplantation of purified autologous bone marrow-derived stem cells and mesenchymal stem cells.

SUMMARY:
This study is a single arm, single center trial to study the safety and efficacy of purified autologous bone marrow derived stem cells and mesenchymal stem cells for the treatment of children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a chronic childhood disorder defined by a range of motor and cognitive impairments and results in a substantial suffering to the patient and a tremendous socio-economic burden to the individual, family, and healthcare system. With no effective treatments or interventions, therapies for CP are currently focused on supportive and management strategies. Stem cell transplantation has been suggested as a putative intervention for neural pathology, as mesenchymal and neural stem cells, as well as olfactory ensheathing glia and Schwann cells, which have shown some regenerative and functional efficacy in experimental central nervous system disorders.

In this trial, the investigators study the safety and efficacy of the intrathecal transplantation of specific populations of purified autologous bone marrow-derived stem cells and mesenchymal stem cells in patients with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Must be more than 2 year of age and less than 12 years of age at the time of screening for inclusion in the study.
* Clinical evidence of a non-progressive motor disability due to brain dysfunction.
* Willing to comply with all study procedures.
* Gross Motor Function Classification Score level II-V

Exclusion Criteria:

Known history of:

* Intractable seizures
* Traumatic brain injury
* Genetic disorder
* Current Infection
* Renal insufficiency
* Hepatic disease
* HIV+ (as demonstrated by positive blood test)
* Immunosuppression
* Infectious related neurological injury
* Other etiologies such as degenerative, mitochondrial, and metabolic disorders
* Normal brain MRI
* Evidence of acute illness such as fever (temperature > 37.5 C), vomiting, diarrhea, wheezing or crackles
* Progressing neurological disease (Batten Disease, Leukodystrophies, Neurotransmitter disorders)
* Microcephaly, macrocephaly, cortical malformations, or genetic disorders of dysgenesis
* Pulmonary disease requiring ventilator support
* Unwillingness to return for follow-up visits
* Contraindications to MRI

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Motor Performance. | 6 months
  GMPM (Gross Motor Performance Measure) as a standard measurement tool for assessing quality of movement.

SECONDARY OUTCOMES:
Motor function studies | 1 year
  Total volumes and specific tract lesions will be studied and correlated with functional outcomes.
Specific white matter tract analysis using MRI | 6 months
  Changes on brain Diffusion Tensor Image (DTI).

IPD SHARING:
Plan to Share IPD: Undecided